CLINICAL TRIAL: NCT01941264
Title: Community-based Scheduled Screening and Treatment of Malaria in Pregnancy for Improved Maternal and Infant Health: a Cluster-randomized Trial in The Gambia, Burkina Faso and Benin
Brief Title: Community-based Screening and Treatment of Malaria in Pregnancy: a Cluster-randomized Trial
Acronym: COSMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Tropical Institute (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Centre Muraz (Other); Imperial College London (Other); World Health Organization (Other); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6800110; ISRCTN37259296 (Registry Identifier: ISRCTN register)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2015-11

CONDITIONS: Malaria, Antepartum; Maternal Malaria During Pregnancy - Baby Not Yet Delivered; Small for Gestational Age (Disorder)
Keywords: malaria; placenta; pregnancy; plasmodium falciparum; screening and treatment; rapid diagnostic test; coartem; artemether-lumefantrine; community health worker
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Therapeutics; Rapid Diagnostic Tests; Artemether, Lumefantrine Drug Combination; Community Health Workers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- community based screening and treatment (Active Comparator): CHWs will identify pregnant women in the village and encourage to go to the antenatal care clinic, furthermore, once a month the community health worker will screen the pregnant women for malaria with a rapid diagnostic test and treat with artemether-lumefantrine in case of a positive test result.
  Interventions: Other: community based screening and treatment
- Control (No Intervention): All pregnant women will be identified in the study area and asked for participation to the study. No intervention will take place.

INTERVENTIONS:
Other: community based screening and treatment — Already described in intervention arm description.
  Other Names: Rapid diagnostic test; Coartem; Artemether-lumefantrine; malaria village worker; village health worker; community case management
  Arms: community based screening and treatment

SUMMARY:
Malaria is a common disease in Africa and a major health problem. Pregnant women are also at risk of malaria. Malaria in pregnancy is life threatening to both the mother and the baby she is carrying. It can result in the destruction of the mother's blood and in babies with a lower birth weight than normal, making them less healthy in their first years of life. These risks are even higher in women having their first pregnancy.

When a woman is pregnant she should go to the Antenatal clinic (ANC) for care. Usually the ANC health staff gives the woman intermittent preventable treatment (IPTp-SP) against malaria. This drug helps protect the woman against getting malaria. Each pregnant woman should receive at least 2 doses of this drug during their pregnancy; thus, they should go the ANC at least 2 times during their pregnancy. However, many women still do not go often to the ANC for health care during their pregnancy.

This study would like to see whether community health workers (CHW) can work with pregnant women to encourage them to attend ANC more often. Also, the CHW will test a pregnant woman every month for malaria with a rapid test. If a woman has malaria, the CHW will treat her in her home instead of the woman having to go a health clinic for treatment. The woman will be treated with a different drug than the drug that is given at the ANC visits. Our hypothesis is that this will improve the care and management of malaria during pregnancy and this will improve the health of women and their newborns. To see whether this strategy improved the health of women and their newborns, we will take a small piece of the placenta at delivery to test for malaria and we will weigh the baby. We will test this strategy in multiple communities. We will compare this to pregnant women in communities where this strategy was not followed, thus where pregnant women received standard care.

Participants will be pregnant women. There are no direct benefits for participating in the study, except the outcome of our research question that is possible health benefits in the intervention group. The drugs involved are tested safe in pregnant women from second trimester on.

DETAILED DESCRIPTION:
Community health workers (CHWs) that will be working in intervention villages will be trained on community-based case management of malaria by monthly testing of pregnant women using a rapid diagnostic test (RDT). They will also be taught the benefit of pregnant women visiting the antenatal clinics (ANC) and that women should receive intermittent preventive treatment with sulphadoxine-pyrimethamine (SP) at the ANC according to WHO guidelines.

The CHWs will try to identify all pregnant women in their villages and encourage them to visit the ANC as early as possible in their pregnancy. The CHW will check after one week if the ANC was visited. For women who do not attend the ANC, the CHW will further encourage and discuss reasons for non-attendance. Subsequently the CHW will visit the woman's house every month to test for malaria with a RDT.The CHW will give a full course of AL to any woman with a positive RDT. The CHW will also collect a blood slide and a blood spot on filter paper for later analysis in the laboratory. The CHWs will return to women who were treated for malaria to check uptake and compliance by using a short questionnaire and checking the empty packaging of the treatment at the end of the course.

In control communities, CHW will not be trained to do RDTs and give AL to pregnant women. The only data collection will occur during ANC visits.

All women are asked to deliver in collaborating health centres. Peripheral blood will be tested for hemoglobin, malaria infection and resistance against SP. A placenta biopsy will be collected and all babies will be weighed and examined.

ELIGIBILITY:
Inclusion Criteria:

* Residence in the study area and intention to stay in the area for the duration of the pregnancy and for delivery.
* Aged at least 16 years (pregnant adolescents younger than 16 years will be considered only if they are accompanied by a responsible adult (in the Gambia) or married (considered an adult by marriage in Burkina Faso and Benin.)
* Willing to provide biological samples as and when required during the study period (blood and placental biopsy)
* Informed consent

Exclusion Criteria:

* A history of sensitivity to sulphonamides.
* Already participating in another research study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4265 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Placental malaria | After delivery
  Placental malaria will be diagnosed by microscopy of placental biopsies and polymerase chain reaction (PCR) on placental blood.

SECONDARY OUTCOMES:
Birth weight | After delivery
  Babies of mothers included in the study will be weighed after delivery.

OTHER OUTCOMES:
antenatal care clinic attendance | Throughout inclusion (+/- 6 months)
  A field worker will identify all eligible pregnant women and will follow-up on ANC attendance through lists at the antenatal care clinic
Resistance to sulphadoxine-pyrimethamine (SP) | At delivery
  Samples infected with P.falciparum will be checked for resistance profile for sulphadoxine-pyrimethamine
Peripheral malaria infection | Throughout inclusion (+/- 6 months)
  Each collected filter paper en microscopy slide (both in antenatal care clinics and from community health worker visits) will be checked for the presence of malaria parasites.
hemoglobin | At delivery
  Peripheral blood sample will be tested for hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Henk Schallig, Dr, Study Director — Royal Tropical Institute (KIT)
Locations (3):
- Centre de Recherches Entomologiques de Cotonou (CREC), Cotonou, Benin
- Clinical Research Unit of Nanoro URCN/CMA, Centre Muraz (CM), Nanoro, Burkina Faso
- Medical Research Council (MRC), Fajara, The Gambia

REFERENCES:
- [Background] Scott S, Mens PF, Tinto H, Nahum A, Ruizendaal E, Pagnoni F, Grietens KP, Kendall L, Bojang K, Schallig H, D'Alessandro U. Community-based scheduled screening and treatment of malaria in pregnancy for improved maternal and infant health in The Gambia, Burkina Faso and Benin: study protocol for a randomized controlled trial. Trials. 2014 Aug 28;15:340. doi: 10.1186/1745-6215-15-340. PMID 25169073
- [Derived] Natama HM, Moncunill G, Vidal M, Rouamba T, Aguilar R, Santano R, Rovira-Vallbona E, Jimenez A, Some MA, Sorgho H, Valea I, Coulibaly-Traore M, Coppel RL, Cavanagh D, Chitnis CE, Beeson JG, Angov E, Dutta S, Gamain B, Izquierdo L, Mens PF, Schallig HDFH, Tinto H, Rosanas-Urgell A, Dobano C. Associations between prenatal malaria exposure, maternal antibodies at birth, and malaria susceptibility during the first year of life in Burkina Faso. Infect Immun. 2023 Oct 17;91(10):e0026823. doi: 10.1128/iai.00268-23. Epub 2023 Sep 27. PMID 37754682
- [Derived] Natama HM, Moncunill G, Rovira-Vallbona E, Sanz H, Sorgho H, Aguilar R, Coulibaly-Traore M, Some MA, Scott S, Valea I, Mens PF, Schallig HDFH, Kestens L, Tinto H, Dobano C, Rosanas-Urgell A. Modulation of innate immune responses at birth by prenatal malaria exposure and association with malaria risk during the first year of life. BMC Med. 2018 Nov 2;16(1):198. doi: 10.1186/s12916-018-1187-3. PMID 30384846
- [Derived] COSMIC Consortium. Community-based Malaria Screening and Treatment for Pregnant Women Receiving Standard Intermittent Preventive Treatment With Sulfadoxine-Pyrimethamine: A Multicenter (The Gambia, Burkina Faso, and Benin) Cluster-randomized Controlled Trial. Clin Infect Dis. 2019 Feb 1;68(4):586-596. doi: 10.1093/cid/ciy522. PMID 29961848